CLINICAL TRIAL: NCT02549131
Title: Cesarean Wound Closure in Women With BMI 40 or Greater: A Randomized Controlled Trial Comparing Subcuticular Suture to Surgical Staples
Brief Title: Cesarean Wound Closure in Women With BMI 40 or Greater
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatrix (Other)
Collaborators: Banner Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Cesarean Closure
Record Dates: First submitted 2015-08-28; First posted 2015-09-15 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: C.Delivery; Penetration, Pregnant Uterus, by Instrument; Obesity
MeSH Terms: conditions — Obesity | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suture (Active Comparator): Randomizing to Suture closure of Cesarean Section wound. In woman meeting inclusion criteria and not meeting exclusion criteria.
  Interventions: Procedure: Randomizing to Suture or Staple closure of Cesarean section
- Staples (Active Comparator): Women in this Arm will be assigned to Standard Surgical Staples closure of Cesarean section.
  Women will have met inclusion criteria and not meet exclusion criteria and willing to consent to study. Intervention is the randomization to either Arm. Both are standard of care at this facility.
  Interventions: Procedure: Randomizing to Suture or Staple closure of Cesarean section

INTERVENTIONS:
Procedure: Randomizing to Suture or Staple closure of Cesarean section — Randomizing to either surgical subcuticular suture or surgical staples in women of BMI greater than 40 undergoing Cesarean section delivery.
  Other Names: suture or staples for skin closure

SUMMARY:
The purpose of this randomized controlled prospective trial is to guide physicians on the most effective evidenced based skin closure during a cesarean section for the obese gravida, defined as a BMI of 40 or greater. The study will compare two closure methods: subcuticular sutures and surgical staples.

DETAILED DESCRIPTION:
The study will screen and attempt to enroll pregnant women admitted to labor and delivery who have a BMI of 40 or greater. The participants will be randomized to receiving skin closure with subcuticular sutures or surgical staples if they undergo cesarean section. Either technique is currently standard of care. Participants who end up undergoing cesarean section will be included in the final data analysis. The participants will be followed for wound complication in the first 6 weeks post operatively. Wound complication will be defined as wound disruption or infection within 6 weeks post operatively.

Design and Project Type This study is a randomized controlled trial. At the study facility, in 2012 and 2013, over 300 cesarean sections were performed each year in women with BMI of 40 or greater. Based on this, the investigators expect the duration of the study to be 2 years. Randomization and data collection will be completed on 420 women.

Description of Intervention Two interventions will be used in this project: subcuticular suture and surgical staples. The subcuticular suture will be the size and type of suture chosen by the surgeon at the time of cesarean. The surgical staples will be the standard staples used on the labor and delivery unit.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* Time to approach and consent the patient prior to undergoing cesarean delivery
* Able to give informed consent, include age 18 or greater and ability to read and understand English
* BMI of 40 or greater on most recent hospital documentation
* Willingness to participate in the study and ability to read, understand and sign the informed consent document

Exclusion Criteria:

* Inability to give informed consent, including inability to read and understand English and age under 18 years
* Evidence of current skin infection or breakdown at or near the site of surgical incision
* Any immune compromised status, including AIDS
* Negative pressure wound therapy applied at time of surgery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 232 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Rate of wound complication, comparing the outcomes from the two arms | 2 years
  Rate of wound complication comparing the outcomes of subcuticular sutures to surgical staples for cesarean wound closure in the obese gravida during the first 6 weeks postpartum.

SECONDARY OUTCOMES:
Frequency of and risk factors for wound complication after cesarean delivery in the obese gravida. | 2 years
  wound complication frequency
Type and location of cesarean incisions in the obese gravida. | 2 years
  type and location of incisions
Effect of medical comorbidities on wound disruption. | 2 years
  medical comorbidities on wound disruption

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Perlow, MD, Principal Investigator — Pediatrix
Locations (2):
- United States (2):
  - Banner University Medical Center - Phoenix, Phoenix, Arizona
  - University of Colorado Denver, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No
no individual patient data will be shared

REFERENCES:
- [Background] Dahlke JD, Mendez-Figueroa H, Rouse DJ, Berghella V, Baxter JK, Chauhan SP. Evidence-based surgery for cesarean delivery: an updated systematic review. Am J Obstet Gynecol. 2013 Oct;209(4):294-306. doi: 10.1016/j.ajog.2013.02.043. Epub 2013 Mar 1. PMID 23467047
- [Background] ACOG practice bulletin no. 105: bariatric surgery and pregnancy. Obstet Gynecol. 2009 Jun;113(6):1405-1413. doi: 10.1097/AOG.0b013e3181ac0544. No abstract available. PMID 19461456
- [Background] Myles TD, Gooch J, Santolaya J. Obesity as an independent risk factor for infectious morbidity in patients who undergo cesarean delivery. Obstet Gynecol. 2002 Nov;100(5 Pt 1):959-64. doi: 10.1016/s0029-7844(02)02323-2. PMID 12423861
- [Background] Alanis MC, Villers MS, Law TL, Steadman EM, Robinson CJ. Complications of cesarean delivery in the massively obese parturient. Am J Obstet Gynecol. 2010 Sep;203(3):271.e1-7. doi: 10.1016/j.ajog.2010.06.049. Epub 2010 Aug 3. PMID 20678746
- [Background] Conner SN, Verticchio JC, Tuuli MG, Odibo AO, Macones GA, Cahill AG. Maternal obesity and risk of postcesarean wound complications. Am J Perinatol. 2014 Apr;31(4):299-304. doi: 10.1055/s-0033-1348402. Epub 2013 Jun 13. PMID 23765707
- [Background] Mackeen AD, Devaraj T, Baxter JK. Cesarean skin closure preferences: a survey of obstetricians. J Matern Fetal Neonatal Med. 2013 May;26(8):753-6. doi: 10.3109/14767058.2012.755509. Epub 2013 Jan 11. PMID 23211124
- [Background] Perencevich EN, Sands KE, Cosgrove SE, Guadagnoli E, Meara E, Platt R. Health and economic impact of surgical site infections diagnosed after hospital discharge. Emerg Infect Dis. 2003 Feb;9(2):196-203. doi: 10.3201/eid0902.020232. PMID 12603990
- [Background] Pevzner L, Swank M, Krepel C, Wing DA, Chan K, Edmiston CE Jr. Effects of maternal obesity on tissue concentrations of prophylactic cefazolin during cesarean delivery. Obstet Gynecol. 2011 Apr;117(4):877-882. doi: 10.1097/AOG.0b013e31820b95e4. PMID 21422859
- [Background] McLean M, Hines R, Polinkovsky M, Stuebe A, Thorp J, Strauss R. Type of skin incision and wound complications in the obese parturient. Am J Perinatol. 2012 Apr;29(4):301-6. doi: 10.1055/s-0031-1295637. Epub 2011 Nov 21. PMID 22105439
- [Background] Thornburg LL, Linder MA, Durie DE, Walker B, Pressman EK, Glantz JC. Risk factors for wound complications in morbidly obese women undergoing primary cesarean delivery. J Matern Fetal Neonatal Med. 2012 Sep;25(9):1544-8. doi: 10.3109/14767058.2011.653422. Epub 2012 Feb 13. PMID 22233403